CLINICAL TRIAL: NCT05942261
Title: Rehabilitation Methods of Children With Cochlear Implant: a Cross-sectional Survey
Brief Title: Rehabilitation Methods of Children With Cochlear Implant
Acronym: MRSI
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, mari Giorgia, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 5685
Record Dates: First submitted 2023-07-04; First posted 2023-07-12 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Deafness Neurosensory
Keywords: cochlear implant; deafness; rehabilitation
MeSH Terms: conditions — Hearing Loss, Sensorineural; Deafness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey to collect data — The study is a survey aimed to collect data about rehabilitation methods

SUMMARY:
The goal of this observational study is to describe the type of the rehabilitation method for italian children with cochlear implant . The main questions are:

What is the most used rehabilitation methods in implanted children? Which is the prevalence of each method related to the clinical features of the patients?

DETAILED DESCRIPTION:
The cochlear implant represents the gold standard in the treatment of children with bilateral severe-profound deafness. However, the current Italian and international guidelines do not address the issue of rehabilitation and how the different rehabilitation methods should be applied in relation to the different clinical pictures. The aim of this study is therefore to describe which methods are used today in the rehabilitation of deaf children with cochlear implants followed at the Phoniatrics and Speech Therapy service of the A. Gemelli Polyclinic Foundation. The creation of a questionnaire directed to the speech therapist who treats the specific patient is available in order to collect data concerning the characteristics of the setting and the rehabilitation method in relation to the most applied methodologies, i.e. Auditory-verbal therapy, oral-cognitive therapy, bimodal method and the Drežančić method.

Inclusion Criteria:

* Children diagnosed with severe-profound hearing loss and cochlear implant carriers followed at the Fondazione Policlinico universitario a. Gemelli in the last 10 years;
* Age >12 months and <10 years

Exclusion Criteria:

* Children diagnosed with mild to moderate hearing loss without a cochlear implant;
* Age <12 months and >10 years

Outcomes measures

* Describe which methods are used today in the rehabilitation of the deaf child with a cochlear implant
* Describe the prevalence of the different methodologies in relation to the clinical characteristics of the patients.

Endpoints:

-% distribution of the 4 rehabilitation methods: cognitive oralism, verb-tonal, Auditory-Verbal therapy and bimodal

- % distribution of the 4 rehabilitation methods: cognitive oralism, verbal-tonal, Auditory-Verbal Therapy and bimodal in relation to the clinical characteristics of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe to profound hearing loss who underwent cochlear implant placement surgery in the last 10 years;
* Age >12 months and <10 years

Exclusion Criteria:

* Patients diagnosed with mild to moderate hearing loss without a cochlear implant
* Age <12 months and >10 years

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with severe-profound hearing loss and cochlear implant carriers followed at the Fondazione Policlinico Universitario A. Gemelli, Rome
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Methods | 3 months
  Describe which methods are used today in the rehabilitation of the deaf child with a cochlear implant.

SECONDARY OUTCOMES:
Prevalence | 2 months
  Describe the prevalence of the different methodologies in relation to the clinical characteristics of the patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli, Roma, RM, Italy